CLINICAL TRIAL: NCT06250569
Title: Application of the Revised Morphological Uterus Sonographic Assessment (MUSA) Criteria to Diagnose Adenomyosis in Fertile Women
Brief Title: Adenomyosis in Fertile Women in MUSA Criteria
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya nour Elzanaty, principal invistigator, Assiut University
Other Study IDs: Adenomyosis in fertile womens
Record Dates: First submitted 2024-01-26; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Adenomyosis
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- first group: women with with adenomyosis
- second group: women without adenomyosis

SUMMARY:
1. To estimate the prevalence of adenomyosis in fertile women aged 18-30 years using the revised MUSA ultrasound criteria.
2. To evaluate clinical risk factors that are associated with adenomyosis diagnosis in this population

DETAILED DESCRIPTION:
Adenomyosis is a benign condition characterized by the presence endometrial glands and stroma within the myometrium. Its prevalence varies from 5-70%. The definitive diagnosis of adenomyosis is based mainly on histological assessment of hysterectomy specimens. This led to a concept that adenomyosis affects only parous women between 35-50 years who complain of dysmenorrhea and heavy menstrual bleeding. Magnetic Resonance Imaging (MRI) can detect adenomyosis with a sensitivity of 80%. Transvaginal ultrasound using the revised Morphological Uterus Sonographic Assessment (MUSA) criteria can detect adenomyosis non-invasively at a lower cost. Such advancements in imaging techniques allow studying the prevalence of the disease in wider range of population including young women.

ELIGIBILITY:
Inclusion Criteria:

* women with regular menstrual cycle attending outpatient clinic for contraception counseling
* age 18 -30 years old

Exclusion Criteria:

* Women on hormonal contraception
* Infertile women
* Associated pathologies like endometriosis, uterine fibroids. and ovarian cysts

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include women with regular menstrual cycle attending outpatient clinic for contraception counseling( age 18 -30 years old ; written consent will be obtained )
Sampling Method: Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
adenomyosis in fertile women | 1.5 year
  Estimation of the prevalence of adenomyosis diagnosed using revised MUSA criteria among fertile women aged 18-30 years.

CONTACTS AND LOCATIONS:
Overall Officials: safwat abdelrady, Prof, Study Director — Assiut University
Locations (1):
- Assuit university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marion LL, Meeks GR. Ectopic pregnancy: History, incidence, epidemiology, and risk factors. Clin Obstet Gynecol. 2012 Jun;55(2):376-86. doi: 10.1097/GRF.0b013e3182516d7b. PMID 22510618
- [Background] Practice Committee of American Society for Reproductive Medicine. Medical treatment of ectopic pregnancy. Fertil Steril. 2008 Nov;90(5 Suppl):S206-12. doi: 10.1016/j.fertnstert.2008.08.049. PMID 19007632
- [Background] Karol D, Williamson M, Pereira N. Successful Expectant Management of a Tubal Ectopic Pregnancy. J Minim Invasive Gynecol. 2024 Feb;31(2):92-94. doi: 10.1016/j.jmig.2023.11.011. Epub 2023 Nov 30. No abstract available. PMID 38042476
- [Background] Harmsen MJ, Van den Bosch T, de Leeuw RA, Dueholm M, Exacoustos C, Valentin L, Hehenkamp WJK, Groenman F, De Bruyn C, Rasmussen C, Lazzeri L, Jokubkiene L, Jurkovic D, Naftalin J, Tellum T, Bourne T, Timmerman D, Huirne JAF. Consensus on revised definitions of Morphological Uterus Sonographic Assessment (MUSA) features of adenomyosis: results of modified Delphi procedure. Ultrasound Obstet Gynecol. 2022 Jul;60(1):118-131. doi: 10.1002/uog.24786. PMID 34587658